CLINICAL TRIAL: NCT05831007
Title: An Open Label Dose Escalation Clinical Trial to Evaluate the Safety and the Efficacy of LX102-C01 in Patients With Neovascular Age-Related Macular Degeneration (nAMD)
Brief Title: Safety and Efficacy Study of LX102-C01 Treatment of Neovascular Age-Related Macular Degeneration (nAMD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Innostellar Biotherapeutics (Unknown)
Responsible Party: Principal Investigator, Xiaodong Sun, PhD, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHGH-LX102-C01
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LX102-C01 Injection (Experimental): Potential doses:
  3E10 vg, 0.06 mL/eye/dose
  1E11 vg, 0.06 mL/eye/dose
  Interventions: Genetic: LX102-C01 Injection

INTERVENTIONS:
Genetic: LX102-C01 Injection — Qualified subjects will receive a single unilateral intravitreal injection of LX102-C01 at Day 0 in the trial.

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of LX102-C01 treatment of nAMD. This study will enroll subjects aged ≥ 50 years old to receive a single unilateral intravitreal (IVT) injection of LX102-C01 to evaluate its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent, and willing to attend follow-up visits.

1. Age ≥ 50
2. Diagnosis of active CNV secondary to neovascular AMD
3. The study eye must have a best-corrected E-ETDRS visual acuity letter score of less than or equal to 63.
4. Subjects must have received a minimum of 2 injections within 6 months prior to screening.
5. Demonstrated a meaningful response to anti-VEGF therapy

Exclusion Criteria:

1. CNV or macular edema in the study eye secondary to diseases other than nAMD
2. Retinal detachment, uveitis, uncontrolled glaucoma in the study eye, or any condition preventing visual acuity improvement
3. Acute coronary syndrome, myocardial infarction or coronary artery revascularization, CVA, TIA in the last 6 months
4. Uncontrolled hypertension defined as average SBP ≥160 mmHg or an average DBP ≥100 mmHg
5. Uncontrolled diabetes defined as HbA1c >7.5%

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 52 weeks
  Incidence of adverse events (AEs) within 52 weeks of LX102-C01 intravitreal injection at different doses
Incidence of serious adverse events (SAEs) | 52 weeks
  Incidence of serious adverse events (SAEs) within 52 weeks of LX102-C01 intravitreal injection at different doses

SECONDARY OUTCOMES:
Mean change in BCVA from Baseline | 24 weeks, 52weeks
  BCVA measured by ETDRS
Mean change in Central Subfield Thickness (CST) from Baseline | 24 weeks, 52 weeks
  To evaluate the effect of LX102-C01 on CST
Mean number of anti-VEGF injections over time | 52 weeks
  Mean number of anti-VEGF injections over time
Change of quality of life scores (VFQ-25) from Baseline | 52 weeks
  Changes of VFQ-25 questionaire from Baseline to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No